CLINICAL TRIAL: NCT04186338
Title: Daily Physical Activity in Children and Adolescents With Low Lumbar and Sacral Level Myelomeningocele
Brief Title: Daily Physical Activity in Myelomeningocele
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Other Study IDs: 09.2017.168
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Physical Activity
Keywords: Activity energy expenditure; Moderate to vigorous physical activity; Myelomeningocele
MeSH Terms: conditions — Motor Activity; Meningomyelocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with myelomeningocele: Patients diagnosed myelomeningocele with the neurological level between L5 and S3
  Interventions: Device: Omnidirectional accelerometer monitor (3x3 cm and 16 g, Actical®, Philips Respironics)
- Healthy controls: age-, sex-, and body mass index-matched healthy controls
  Interventions: Device: Omnidirectional accelerometer monitor (3x3 cm and 16 g, Actical®, Philips Respironics)

INTERVENTIONS:
Device: Omnidirectional accelerometer monitor (3x3 cm and 16 g, Actical®, Philips Respironics) — All participants were instructed to wear monitors for five consecutive days except during water-based activities. Data for each participant was collected to ensure included three valid weekdays. Daily activity energy expenditure (kcal/kg/min), and sedentary, light, moderate and vigorous levels (min) were examined using a software program.

SUMMARY:
Obesity is getting more common and challenging to treat in children and adolescents with myelomeningocele. Therefore, it is becoming more important to determine daily physical activity in these patients. Daily walking performance and average steps per day in patients with low lumbar and sacral level myelomeningocele are shown to not differ from healthy controls. Step counts can not reflect all torsional accelerations associated with daily living activities. Omnidirectional accelerometers provide all types of body movement outputs and give detailed parameters of physical activity level and energy expenditure. There is no data about energy expenditure and physical activity level of the patients with myelomeningocele in daily routine. This study aims to quantify energy expenditure and physical activity of children and adolescents with low lumbar and sacral level myelomeningocele.

DETAILED DESCRIPTION:
Children and adolescents with low lumbar and sacral level myelomeningocele, and age-, sex-, and BMI-matched controls were included. Omnidirectional accelerometer monitor (Actical®) was used to assess activity energy expenditure and daily durations spent in sedentary, light activity and moderate to vigorous physical activity (MVPA).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed myelomeningocele with the neurological level between L5 and S3
* Patients aged between 6 and 16 years
* Independent ambulatory patients without an assistive device or braces

Exclusion Criteria:

* Presence of disorders other than myelomeningocele that affect physical activity or exercise (e.g. rheumatic disease, cardiovascular disease)
* Unable to wear omnidirectional accelerometer monitor (Actical®, Philips Respironics) for five consecutive days

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents with low lumbar and sacral level myelomeningocele and their age-, sex-, and body mass index (BMI)-matched healthy peers were included.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Average Activity energy expenditure (AEE) | After wearing monitors for five consecutive days
  Activity energy expenditure (AEE) (kcal/kg/min) refers to thermogenesis from all activities associated with daily living. An average amount of three valid weekdays will be calculated.

SECONDARY OUTCOMES:
Average physical activity durations | After wearing monitors for five consecutive days
  The sedentary level (min) is the total amount of time when AEE below 0.01 kcal/kg/min. The light level is the total amount of time when AEE between 0.01 and 0.04 kcal/kg/min. The moderate level is the total amount of time when AEE between 0.04 and 0.10 kcal/kg/min. The vigorous level (min) is the total amount of time when AEE above 0.10 kcal/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Kardelen Gencer Atalay, Principal Investigator — Marmara University

REFERENCES:
- [Derived] Gencer-Atalay K, Karadag-Saygi E, Uzuncakmak B, Keskin A, Furtun Y, Guven H, Uzunoglu I, Kurtel H. Daily Physical Activity in Children and Adolescents with Low Lumbar and Sacral Level Myelomeningocele. Dev Neurorehabil. 2021 Apr;24(3):145-149. doi: 10.1080/17518423.2020.1800855. Epub 2020 Aug 4. PMID 32748658